CLINICAL TRIAL: NCT03071185
Title: The Efficacy and Safety of Lower Limb Nerve Blocks in Postoperative Analgesia for the Free Flap Donor Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xia Zhang (Other)
Responsible Party: Sponsor-Investigator, Xia Zhang, Associate Professor, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ChinaMedicalU
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Elective Reconstructive Surgery; Pain, Post Operative
Keywords: free flap; nerve block; elective reconstructive surgery; dexmedetomidine; anterolateral thigh flaps
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group PCA+B (Experimental): Both intravenous PCA and lower limb blocks were used. For patients with fibular flaps harvested, femoral nerve block and common peroneal nerve block with ropivacaine were administered. For patients with ALT flaps harvested, femoral nerve block with ropivacaine was administered.The interventions are femoral nerve block, common peroneal nerve block.
  Interventions: Procedure: femoral nerve block, common peroneal nerve block
- Group PCA (No Intervention): Only intravenous patient controlled analgesia (PCA) was used postoperatively.
- Group PCA+B+D (Experimental): Both intravenous PCA and lower limb blocks with dexmedetomidine as additivewere used.
  Interventions: Procedure: femoral nerve block, common peroneal nerve block

INTERVENTIONS:
Procedure: femoral nerve block, common peroneal nerve block — For patients with fibular flaps harvested, femoral nerve block and common peroneal nerve with ropivacaine were administered. For patients with ALT flaps harvested, femoral nerve block with ropivacaine was administered.
  Other Names: lower limb blocks with dexmedetomidine as additivewere
  Arms: Group PCA+B; Group PCA+B+D

SUMMARY:
The use of free fibular flaps and anterolateral thigh (ALT) flaps for repairing the oromandibular defects is well established, whereas few attentions were focused on postoperative analgesia for the donor area. Dexmedetomidine is a more selective and shorter-acting α2 adrenergic receptor. The purpose of this trial is to determine if using lower limb nerve blocks in patients undergoing free flap-based oromandibular reconstruction can significantly decrease use of pain medications and to evaluate the safety of lower limb nerve blocks. We also investigated the effect of adding dexmedetomidine as additive in femoral nerve blocks for postoperative analgesia.

Patients with oromandibular defects who were scheduled for elective reconstructive surgery using free fibular or ALT flaps, were divided into three groups in a randomized, single-blind fashion. In Group PCA, only intravenous patient controlled analgesia (PCA) was used postoperatively. In Group PCA+B, both intravenous PCA and lower limb blocks were used. In Group PCA+B+D, both intravenous PCA and lower limb blocks with dexmedetomidine as additivewere used. Post-operative narcotic usage, post-operative pain score, post-operative anti-emetic usage, vital signs, onset and duration of sensory and motor block, the presence of adverse effects such as nausea and vomiting were recorded.

DETAILED DESCRIPTION:
The use of free fibular flaps and anterolateral thigh (ALT) flaps for repairing the oromandibular defects is well established, whereas few attentions were focused on postoperative analgesia for the donor area. Conventional postoperative pain management following oromandibular reconstruction consists of systemic opioids, which can cause nausea, vomiting, pruritus, urinary retention, constipation and respiratory depression. Adequate postoperative analgesia decreases the incidence of cardiopulmonary complications. Peripheral nerve blocks can attenuate the sensory innervations.The purpose of this trial is to determine if using lower limb nerve blocks in patients undergoing free flap-based oromandibular reconstruction can significantly decrease use of pain medications and to evaluate the safety of lower limb nerve blocks.

Patients with oromandibular defects, who were scheduled for elective reconstructive surgery using free fibular or ALT flaps, were divided into three groups in a randomized, single-blind fashion. In Group PCA, only intravenous patient controlled analgesia (PCA) was used postoperatively. In Group PCA+B, both intravenous PCA and lower limb blocks were used.In Group PCA+B+D, both intravenous PCA and lower limb blocks with dexmedetomidine as additivewere used. For patients with fibular flaps harvested, femoral nerve block and common peroneal nerve with ropivacaine were administered. For patients with ALT flaps harvested, femoral nerve block with ropivacaine was administered. Post-operative narcotic usage, post-operative pain score, post-operative anti-emetic usage, vital signs, onset and duration of sensory and motor block, the presence of adverse effects such as nausea and vomiting were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis or presumed diagnosis of oral and maxillofacial tumor.
* Undergoing microsurgical oromandibular reconstruction with free fibular flaps and anterolateral thigh flaps.
* Greater than 18 years old.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* True allergy to local anesthetics or opioids.
* History of addiction to narcotics within the last 24 months
* History of chronic pain on opioids within the last 24 months.
* Specific mental health issues such as schizophrenia or bipolar disorder.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Post-operative Narcotic Usage | 48 hours
  Total intravenous sulfentanyl usage for rescue analgesia in first 48 hours post-operatively after free fibular flaps and anterolateral thigh flap reconstruction.
duration of sensory blockade | 48 hours
  the time of sensory recovery
duration of motor blockade | 48 hours
  the time of motor recovery
onset of sensory blockade | 48 hours
  the time to sensory blockade
onset of motor blockade | 48 hours
  the time to motor blockade

SECONDARY OUTCOMES:
Post-operative Anti-emetic Usage | 48 hours
  Post-operative Anti-emetic Usage is defined as the total amount of IV tropisetron administered to a patient during the first 48 hours post-operatively.
vital signs | 48 hours
  hear rate, blood pressure, SPO2
Post-operative Pain Score | 48 hours
  Post-operative Pain Score is defined using Visual Analog Scale (VAS), a patient reported pain score on a scale of 0-10.
adverse effects | 48 hours
  such as bradycardia, hypotension,respiratory depression, postoperative sedation

CONTACTS AND LOCATIONS:
Overall Officials: xia zhang, Ph.D,MD, Principal Investigator — School & Hospital of Stomatology, China Medical University, China
Locations (1):
- School & Hospital of Stomatology, China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No